CLINICAL TRIAL: NCT05964803
Title: Males Living With HIV and LUTS: A Case-control Study.
Brief Title: Lower Urinary Tract Symptoms in Males Living With HIV
Status: Completed | Type: Observational
Sponsor: Koç University (Other)
Responsible Party: Principal Investigator, Ersin Köseoglu, MD, Koç University
Other Study IDs: KocUrol5
Record Dates: First submitted 2023-07-09; First posted 2023-07-28 (Actual); Last update posted 2024-04-17 (Actual); Status verified 2024-04

CONDITIONS: HIV Seropositivity; Lower Urinary Tract Symptoms
MeSH Terms: conditions — HIV Seropositivity; Lower Urinary Tract Symptoms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Males living with HIV: Males living with HIV and followed by infectious diseases clinic will be directed to Urology department.
  Interventions: Diagnostic Test: Questionnaires
- HIV-negative controls: Males admitted to Infectious Diseases clinic and documented to be HIV-negative.
  Interventions: Diagnostic Test: Questionnaires

INTERVENTIONS:
Diagnostic Test: Questionnaires — MLWH and control groups were asked to complete the following questionnaires: International Consultation on Incontinence Questionnaire - Male Lower Urinary Tract Symptoms (ICIQ-MLUTS), ICIQ-Short Form (ICIQ-SF), International Prostate Symptom Score (IPSS), King's Healthcare Questionnaire (KHQ), 8-item Overactive Bladder Questionnaire (OAB-V8), Urogenital Distress Inventory 6 and 7 (UDI 6 and UDI 7).

SUMMARY:
The primary aim of this study is to learn whether the frequency of lower urinary tract symptoms differ between the males with seronegativity for HIV and males living with HIV.

ELIGIBILITY:
Inclusion Criteria:

* Patients above 18 years old

Exclusion Criteria:

* Non-Turkish speakers
* Previous surgeries or medications for lower urinary tract symptoms

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Males above 18 years old
Study Population: Patients admitted to Infectious Diseases Clinic (100 living with HIV, 100 HIV-negative males) will be directed to Urology clinic. The same questionnaires will be given and scores will be compared.
Sampling Method: Non-Probability Sample
Enrollment: 55 (Actual)
Dates: Start 2023-08-01 (Actual); Primary Completion 2023-12-01 (Actual); Study Completion 2024-01-01 (Actual)

PRIMARY OUTCOMES:
Questionnaire 1 | Day 1
  International Consultation on Incontinence Questionnaire
Questionnaire 2 | Day 1
  Male Lower Urinary Tract Symptoms (ICIQ-MLUTS)
Questionnaire 3 | Day 1
  ICIQ-Short Form (ICIQ-SF)
Questionnaire 4 | Day 1
  International Prostate Symptom Score (IPSS)
Questionnaire 5 | Day 1
  King's Healthcare Questionnaire (KHQ)
Questionnaire 6 | Day 1
  8-item Overactive Bladder Questionnaire (OAB-V8)
Questionnaire 7 | Day 1
  Urogenital Distress Inventory 6 and 7 (UDI 6 and UDI 7).

CONTACTS AND LOCATIONS:
Locations (1):
- Koc University Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No